CLINICAL TRIAL: NCT05729425
Title: Microvessel Ultrasound Imaging of Cutaneous Angiosarcoma
Brief Title: Evaluating the Accuracy of Microvessel Ultrasound Imaging for Detecting Extent of Disease in Patients With Angiosarcoma of the Skin
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit participants due to rare disease
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 21-005183; NCI-2022-09609 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-005183 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2023-02-08; First posted 2023-02-15 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Skin Angiosarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Observational (microvessel ultrasound imaging): Patients undergo microvessel ultrasound imaging on study.
  Interventions: Device: Ultrasound Microvessel Imaging

INTERVENTIONS:
Device: Ultrasound Microvessel Imaging — Undergo microvessel ultrasound imaging
  Other Names: 3D Ultrasound Microvessel Imaging; UMI

SUMMARY:
This study evaluates the accuracy of a new ultrasound technology called microvessel imaging for detecting the extent of disease among patients with angiosarcoma of the skin. Microvessel ultrasound imaging uses high frequency waves to visualize vessels in the skin that are not easily seen using other imaging tests.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the accuracy of depicting extent of disease of cutaneous angiosarcoma before and after neoadjuvant treatment compared to clinical photographs, magnetic resonance imaging (MR) or positron emission tomography (PET)/computed tomography (CT) imaging and surgical pathology both on skin biopsies and surgical excision.

OUTLINE:

Patients undergo microvessel ultrasound imaging on study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Diagnosed with cutaneous angiosarcoma of the breast or scalp and scheduled for trimodality therapy
* Twenty one years of age or older

Exclusion Criteria:

* Unwilling to consent to microvessel ultrasound imaging
* Younger than 21 years of age

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 21 with new diagnosis of cutaneous angiosarcoma of the breast or scalp.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of microvessel ultrasound imaging | Through to study completion up to one year
  Accuracy with respect to gold standard quantitative measures of disease extent and imaging-based measurements will be evaluated using Lin's concordance correlation coefficient along with 95% confidence intervals (CI's). These will be performed separately pre- and post-treatment. Pearson correlations and 95% CI's between imaging modality measurements will also be estimated to help guide future comparative analyses. Bland-Altman plots will also be generated to visualize agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany M Sae-Kho, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials